CLINICAL TRIAL: NCT01046084
Title: A Relative Bioavailability Replicated Crossover Study of Lansoprazole 30 mg Delayed-Release Capsules Under Non-Fasting Conditions.
Brief Title: Lansoprazole 30 mg DR Capsule Replicate Food Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B036522
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Results first posted 2010-03-19 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Lansoprazole

ARMS (2):
- Investigational Test Product (Experimental): Lansoprazole 30 mg Delayed-Release Capsule
  Interventions: Drug: Lansoprazole
- Reference Listed Drug (Active Comparator): Prevacid® 30 mg Delayed-Release Capsule
  Interventions: Drug: Prevacid®

INTERVENTIONS:
Drug: Lansoprazole — 30 mg Delayed-Release Capsule
  Arms: Investigational Test Product
Drug: Prevacid® — 30 mg Delayed-Release Capsule
  Other Names: Lansoprazole (generic name)
  Arms: Reference Listed Drug

SUMMARY:
The object of this study is to compare the relative bioavailability of lansoprazole 30 mg delayed-release capsules (manufactured by TEVA Pharmaceutical Industries, Ltd. and distributed by TEVA Pharmaceuticals USA) with that of PREVACID® capsules (TAP Pharmaceuticals, Inc.) in healthy, adult, subjects under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Body Mass Index of 30 or less
* Males or non-pregnant females
* Normal clinical laboratory test results

Exclusion Criteria:

* Subjects with a significant history of chronic alcohol consumption (past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic, or cardiovascular disease, tuberculosis, epilepsy, asthma (past 5 years), diabetes, psychosis or glaucoma will not be eligible for the study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested will be excluded from the study.
* Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least 30 days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within 30 days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allow to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Female subjects who have used hormonal oral contraceptives within 180 days of dosing will not be allowed to participate.
* Female subjects with a positive or inconclusive pregnancy test result will be withdrawn from the study.
* Subjects who do not tolerate venipuncture will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Parham, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Lansoprazole) First: 30 mg Lansoprazole Delayed-Release Capsules test product dosed in first and third periods followed by 500 mg Prevacid® Capsules reference product dosed in the second and fourth periods.
- Reference (Prevacid®) First: 30 mg Prevacid® Capsules reference product dosed in first and third periods followed by 30 mg Lansoprazole Capsules test product dosed in the second and fourth periods.
Period: First Intervention
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: First Washout of 7 Days
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Washout of 7 Days
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Third Intervention
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Third Washout of 7 Days
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First
Started | 25 | 25
Completed | 23 | 25
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Fourth Intervention
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First
Started | 23 | 25
Completed | 23 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Lansoprazole) First | Reference (Prevacid®) First | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 15 | 10 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Black | 6 | 5 | 11
  Caucasian | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 14 hour period.
Population: All participants that completed the study had their samples analyzed. Replicate study design allowed for 2 sets of samples per subject per treatment (N=96 for both test and reference).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Lansoprazole): 30 mg Lansoprazole Delayed-Release Capsules test product dosed in any period.
- Reference (Prevacid®): 30 mg Prevacid® Capsules reference product dosed in any period.
Arm/Group | Test (Lansoprazole) | Reference (Prevacid®)
Number analyzed (Participants) | 96 | 96
ng/mL | 272.038 (231.03) | 238.043 (175.201)
Statistical Analysis 1: Comparison: Test (Lansoprazole) vs Reference (Prevacid®); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 103, 90% CI 2-sided [86.5 to 123] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 14 hour period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Lansoprazole) | Reference (Prevacid®)
Number analyzed (Participants) | 96 | 96
ng*h/mL | 979.389 (972.74) | 890.06 (780.912)
Statistical Analysis 1: Comparison: Test (Lansoprazole) vs Reference (Prevacid®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 104, 90% CI 2-sided [89.3 to 120] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 14 hour period.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Lansoprazole) | Reference (Prevacid®)
Number analyzed (Participants) | 96 | 96
ng*h/mL | 1060.923 (1066.033) | 938.857 (839.984)
Statistical Analysis 1: Comparison: Test (Lansoprazole) vs Reference (Prevacid®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 107, 90% CI 2-sided [92.5 to 123] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 4 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Test (Lansoprazole) | Reference (Prevacid®)
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 5/50 | 5/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Lansoprazole) (N=50) | Reference (Prevacid®) (N=50)
Headache (General disorders) | 5 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.